CLINICAL TRIAL: NCT04593719
Title: Effect of Lactation Management Model on Breastfeeding Process After Cesarean
Brief Title: Effect of Lactation Management Model on Breastfeeding Process
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Aslı EKER, Lecturer Doctor, Mersin University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Lactation-Management-Model
Record Dates: First submitted 2020-10-06; First posted 2020-10-20 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Lactation; Breastfeeding; Cesarean Section
Keywords: Cesarean section; Breastfeeding; Mother milk; Lactation management model; Breastfeeding training
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experiment (Experimental): Lactation management model is applied to the experimental group.
  Interventions: Other: Experiment
- Control (No Intervention): Lactation management model is not applied to the control group.

INTERVENTIONS:
Other: Experiment — The main components of the Lactation Management Model; breastfeeding training in the prenatal period (from the 30th week of pregnancy), early postpartum period (first 48 hours) skin to skin contact, early breastfeeding, relaxation using a dreaming technique, warm application to the breast, breast massage and for the first 48 hours after postpartum 6 months of continuous support (face to face, by phone, via social media).
  Arms: Experiment

SUMMARY:
Background: While caesarean sections are increasing, breast-feeding rates are decreasing. It is important to implement supportive programs to ensure mothers breast feed for the desired period and infants are fed by only mother's milk.

Aim: In the research, it was aimed to evaluate the effects of lactation management models on mothers' breastfeeding process following a caesarean section.

Methods: The research was conducted as a randomized controlled study and experimentally. Before implementation, Lactation Management Model was developed. Data collection was performed during gestation, first day after postpartum, pre-discharge, on 9th day in face to face interview and in the form of monthly phone interviews up to 6 months. While the experimental group exercised lactation management model, control group received routine lactation practices in clinic.

Conclusions: Among the females in the experimental group, it was found that breastfeeding self-efficacy were higher, and breastfeeding techniques were accurate and successful and breastfeeding only and continuity rates were higher while breastfeeding related breast problems developed less frequently. Lactation management model should be used and expanded to increase breastfeeding rates.

Keywords: Cesarean section, breastfeeding, mother milk, lactation management model, breastfeeding training

DETAILED DESCRIPTION:
It is a birth right of babies to be breast fed and nursed. However, approximately 7.6 million babies cannot be fed with breast milk in the world every year. United Nations International Children's Emergency Fund (UNICEF) declared in its statement that, breast milk access is decreased as household income increases and in nations with high income 1 out of every 5 babies and for low or middle income nations 1 of every 25 babies never fed breast milk (UNICEF, 2018). Worldwide, among the infants under six months old, 40% is fed with breast milk only (UNICEF, 2017). According to Turkey Demographic and Health Survey data, it is found that in Turkey; breast milk feeding rate of infants under 6 months is 41% and in average breast milk feeding period is 1.8 months (TNSA, 2018).

There are many factors affecting whether an infant is breastfed. Delivery method is among one of them. While in OECD nations and in UNITED STATES OF AMERICA 32% of every delivery was caesarean (Health İndicators, 2018; ACOG, 2019), in Turkey this rate is indicated as 52% (TNSA, 2018). Caesarean delivery compared to vaginal delivery is negatively affecting the initial lactation period, milk production and suckling instinct of the infant (Hobbs et al., 2016). Esencan et al. has determined that 42.4% of women who had spinal-caesarean deliveries did not breast feed (Esencan et al., 2018).

Numerous factors are in effect for suckling and milk production. Various studies are performed in the literature it is emphasized that in order to stimulate and increase the milk production; apart from evidence based applications, breast stimulation and other techniques to cure nursing problems should be employed (Anderson et al., 2016). Becker et al. In their systematical compositions; determined that actions such as; resting, music, applying warmth to breast area, massaging, pump aided stimulations increased milk production clinically in a significant manner (Becker et al., 2016). Although applying warmth to breast area, massaging and relaxations techniques for increasing milk production and ensuring long term breast feeding are evidently lacking in the international manuals; early nursing, skin-to-skin contact together with education and support is stated to be positively affecting breast feeding (WHO, 2017; NICE, 2015). Despite all these actions taken national and international breast feeding data still is not at a favorable level. Because initiation of lactation contuniuty and increase in the period of breastfeeding depends on many factors. Education of mother starting from gestational period; care, support and consultancy services should be provided during pregnancy, birth and postpartum periods. This study has been planned in consideriation with the need for a model that includes all this service, maintenance and support, no similar study has been found in the literature that has all these components together.

ELIGIBILITY:
Inclusion Criteria:

* to be between 18-35 years old,
* being in the 30th week of pregnancy,
* 36th week or above with planned caesarean delivery,

Exclusion Criteria:

* risky pregnancy (multiple gestation, Preeclampsia etc.),
* breast operation history,
* health issues of mother or baby that may affect breast feeding process,
* medication use that may affect milk production,
* communication problems related to language,
* failure to be reached via phone after discharge

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women were chosen as it was a study related to breast milk and breastfeeding.
Enrollment: 66 (Actual)
Dates: Start 2017-11-11 (Actual); Primary Completion 2018-07-18 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Continuation of Breastfeeding and Only Breast Milk | 6 month
  Women who are applied lactation management model feed their babies with only breast milk at a higher rate (Measured using Breastfeeding and breastmilk monitoring form.It is a form developed by the researcher, consisting of 4 open-ended questions for the purpose of continuing breastfeeding and breastfeeding and determining additional nutrients other than breast milk).
Breastfeeding Observation Form Scores at Postpartum in The First 48 Hours | The First 48 Hours
  It was determined that women who were applied the Lactation Management Model were able to breastfeed successfully with the appropriate technique (Measured using the Breastfeeding observation form. developed by Armstrong form consists of 25 parameters under 5 main titles. For each parameter, "Percentage of Success" is calculated by taking the frequencies of 0, 1 and 2 scores. "Successful Technique" is indicated as between 46-50 points and "Insufficient Technique" as 45 and below).

SECONDARY OUTCOMES:
Latch Scale Scores and Breast Nipple-Related Discomfort Levels Related to Breastfeeding | First 9 days
  It was found that problems related to the nipple develop less in women who were applied lactation management model (Measured using A breastfeeding charting system and documentation tool. Developed by Jensen et al. scale consists of 5 assessment criteria. Each item has a score of between 0 and 2, and highest score is 10).
Breastfeeding Self-Efficacy Scale Scores | 2 month
  Breastfeeding self-efficacy was higher in women who were applied the Lactation Management Model (Measured using Breastfeeding Self-Efficacy Scale Scores. It was developed by Dennis and is a 5-point Likert type scale. Minimum 14 points and maximum 70 points can be obtained from the scale. A higher score indicates that an increase in breastfeeding self-efficacy).

CONTACTS AND LOCATIONS:
Overall Officials: Aslı EKER, Principal Investigator — Mersin University
Locations (1):
- Mersin University, Yenişehir, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anderson L, Kynoch K, Kildea S. Effectiveness of breast massage in the treatment of women with breastfeeding problems: a systematic review protocol. JBI Database System Rev Implement Rep. 2016 Aug;14(8):19-25. doi: 10.11124/JBISRIR-2016-003058. PMID 27635741
- [Background] ACOG Committee Opinion No. 761: Cesarean Delivery on Maternal Request. Obstet Gynecol. 2019 Jan;133(1):e73-e77. doi: 10.1097/AOG.0000000000003006. PMID 30575678
- [Background] Becker GE, Smith HA, Cooney F. Methods of milk expression for lactating women. Cochrane Database Syst Rev. 2016 Sep 29;9(9):CD006170. doi: 10.1002/14651858.CD006170.pub5. PMID 27684560
- [Background] Esencan YT, et al. Type of delivery, time of ınitial breastfeeding, and skin-to-skin contact of pregnant women participating in childbirth preparation education. Florence Nightingale Journal of Nursing 2018; 26(1): 31-43.
- [Background] Hobbs AJ, Mannion CA, McDonald SW, Brockway M, Tough SC. The impact of caesarean section on breastfeeding initiation, duration and difficulties in the first four months postpartum. BMC Pregnancy Childbirth. 2016 Apr 26;16:90. doi: 10.1186/s12884-016-0876-1. PMID 27118118
- [Derived] Eker A, Aslan E. Effect of Lactation Management Model on Breastfeeding Process After Cesarean: A Prospective Randomized Controlled Study. Reprod Sci. 2024 Apr;31(4):1108-1116. doi: 10.1007/s43032-023-01409-3. Epub 2023 Dec 14. PMID 38097898
- See also: UNİCEF For Every Child, Breastfeeding A Mother's Gift, for Every Child 2018 — http://data.unicef.org/wp-content/uploads/2018/05/180509_Breastfeeding.pdf
- See also: WHO, Protecting, promoting and supporting breastfeeding in facilities providing maternity and newborn services guideline 2017 — http://apps.who.int/iris/bitstream/handle/10665/259386/9789241550086-eng.pdf?sequence=1
- See also: NİCE. Postnatal care up to 8 weeks after birth clinical guideline 37 — http://www.nice.org.uk/guidance/cg37
- See also: Health Indicators — http://khgmozellikli.saglik.gov.tr/svg/inc/saglik_gostergeleri.pdf